CLINICAL TRIAL: NCT01086956
Title: Effect of Adding Sufentanil to Epidural Ropivacaine on Perioperative Metabolic and Stress Responses in Combined General/Epidural Anaesthesia for Geriatric Radical Retropubic Prostatectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Kil Hae Keum, Yonsei University College of Medicine, Seoul, Republic of Korea
Allocation: Randomized | Purpose: Diagnostic
Other Study IDs: 4-2008-0319
Record Dates: First submitted 2010-03-12; First posted 2010-03-15 (Estimated); Last update posted 2010-11-11 (Estimated); Status verified 2010-11

CONDITIONS: Prostatic Cancer
Keywords: patients of prostatic cancer aged more than 65 years
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Ropivacaine; Sufentanil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: epidural infusion of saline, ropivecaine, or ropivacaine and sufentanil

SUMMARY:
The purpose of this study is to compare metabolic and stress responses in combined general/epidural anesthesia in geriatric cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* elective RRP for prostatic cancer scheduled in the morning (9-11 a.m.)
* patients aged more than 65 years
* ASA physical status I or II
* absence of contraindications to epidural approach
* absence of a history of chronic pain or opioid medication

Exclusion Criteria:

* contraindication to epidural catheterization

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
plasma glucose, insulin, cortisol, epinephrine, norepinephrine, prolactin | from preoperative baseline to postoperative 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Hong JY, Yang SC, Yi J, Kil HK. Epidural ropivacaine and sufentanil and the perioperative stress response after a radical retropubic prostatectomy. Acta Anaesthesiol Scand. 2011 Mar;55(3):282-9. doi: 10.1111/j.1399-6576.2010.02360.x. Epub 2010 Nov 25. PMID 21108620